CLINICAL TRIAL: NCT06170229
Title: Comparative Effectiveness of High-intensity Aerobic Exercise and Biomechanical Neuromuscular Exercise for Treatment of Knee Osteoarthritis: a Randomised Open Label Trial
Brief Title: Aerobic Vs Neuromuscular Exercise for Knee OA
Acronym: CANO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT-2023-DK-3
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education and High Intensity Interval Training (eHIIT) (Active Comparator): 1 educational session lasting 1 hour. 12 weeks of supervised High Intensity Interval Training (HIIT) 3 times/week.
  Interventions: Behavioral: eHIIT
- Neuromuscular exercise and education program (NEMEX-e) (Active Comparator): 2 educational sessions lasting 1 hour each. 8 weeks of supervised Neuromuscular Exercise 2 times/week.
  Interventions: Behavioral: NEMEX-e

INTERVENTIONS:
Behavioral: eHIIT — Education and High intensity Interval Training (Aerobic Exercise)
  The focus of the one educational session is rationale for aerobic exercise, expected physiological effects of aerobic exercise, diet when performing an exercise program, how the knee accommodates to exercise (including potential experience of muscle soreness and how that is different from joint pain), and management of potential knee OA symptom flares.
  HIIT is an aerobic exercise form. The eHITT protocol consist of eight 2-minute intervals of high intensity training (with the goal to train at a heart rate of at least 80% of HRmax) followed by 2 minutes of moderate training intensity (with the goal to train at a heart rate of at least 60% of HRmax).
  There will be several types of exercise modalities for aerobic exercise available (treadmills, cross-trainers, row- and cycle ergometers) and participants may choose whichever they prefer.
  Arms: Education and High Intensity Interval Training (eHIIT)
Behavioral: NEMEX-e — Education and Neuromuscular Exercise
  The focus of the two educational sessions is on providing knowledge of OA and treatment options to the participants, with a special focus on knee OA, diet, and exercise and its benefits. Furthermore, advice about self-management is given.
  The exercises are based on neuromuscular principles to improve sensorimotor control and achieve compensatory functional stability. Sensorimotor control is the ability to coordinate muscle activity and maintain functional stability during movement allowing for joint stability during physical activity. Various positions (sitting, lying, standing) are used to achieve the desired postural activity. The overall goal is to obtain muscle control and stability in situations resembling daily life and/or more strenuous activities. The focus is on achieving good quality of the performance in each exercise with appropriate postural orientation (e.g., joint positioned appropriately in relation to each other).
  Arms: Neuromuscular exercise and education program (NEMEX-e)

SUMMARY:
The study aims to compare the effects of an education and High Intensity Interval Training program (eHIIT) with the widely used Neuromuscular Exercise and education program (NEMEX-e) on knee OA symptoms and risk factors for cardiovascular disease in people with knee OA and at least one risk factor for developement of cardiovascular disease. The main research questions the study aims to answer are:

* Is the eHIIT program better than the NEMEX-e program for reducing the risk of cardiovascular disease?
* Are the two programs equally good at providing improvement in knee symptoms?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18- years
* Diagnosis of tibiofemoral knee OA according to the American College of Rheumatology criteria
* Radiographically confirmed diagnosis of tibiofemoral OA based on radiographs not older than 6 months.
* Average knee pain level ≥ 4 (0=No pain and 10=Worst pain) over the past week (7 days)
* At least one of following risk factors for development of cardiovascular disease:

  * Body mass index ≥ 30 kg/m2
  * Hypertension (or in treatment of): Systolic ≥ 135 and/or diastolic ≥ 85 mm Hg
  * Elevated HbA1c (or in treatment of): ≥ 130.7 mg/dL (44 mmol/mol)
  * Elevated Triglycerides (or in treatment of): ≥ 150 mg/dL (1.7 mmol/L)
  * Elevated Cholesterol (or in treatment of) (Low density lipides, LDL): LDL ≥ 54 mg/dL (3.0 mmol/L)

Exclusion Criteria:

* Contraindication to exercise (e.g., resting systolic blood pressure > 200 or diastolic blood pressure > 115, acute or reoccurring chest pain)
* Unstable body weight the last 3 months (gain/loss outside +/- 5 kg)
* Planned weight loss (non-pharmacological, pharmacological, and surgical) during study participation
* Known current cancer
* Major cardiovascular event within the last 5 years
* Insulin dependent type 1 or type 2 diabetes
* Psoriatic, rheumatoid, or gouty arthritis disease
* Generalized pain syndromes such as fibromyalgia
* Lumbar or cervical nerve root compression syndromes
* Scheduled surgery during study participation
* Treatment with biological medication
* Impairments that prevent performance in high intensity aerobic exercise
* Current or planned participation in other health research intervention studies
* Pregnant/considering pregnancy
* Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as a large knee joint effusion, uncontrolled diabetes/hypertension, psychiatric or cognitive disorders, language barriers, or opiate dependency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2max) | Baseline and Week 12
  Cardiopulmonary exercise test (CPET) on an ergometer bicycle for evaluation maximal oxygen consumption (VO2max) measured in ml/min/kg
Knee pain | Baseline and Week 12
  The Knee injury and Osteoarthritis Outcome Score (KOOS) pain subscale (KOOS-pain), a disease-specific patient-reported instrument designed to assess knee pain in patients with knee osteoarthritis.
  The KOOS-pain subscale is scored on a 0-100 scale with 100 indicating no pain and 0 indicating extreme pain.

SECONDARY OUTCOMES:
Maximal oxygen consumption (VO2max) | Week 8 and week 26
  Cardiopulmonary exercise test (CPET) on an ergometer bicycle for evaluation maximal oxygen consumption (VO2max) measured in ml/min/kg
Knee pain | Week 8 and week 26
  The Knee injury and Osteoarthritis Outcome Score (KOOS) pain subscale (KOOS-pain), a disease-specific patient-reported instrument designed to assess knee pain in patients with knee osteoarthritis.
  The KOOS-pain subscale is scored on a 0-100 scale with 100 indicating no pain and 0 indicating extreme pain.
Body Mass | Baseline, Week 12 and Week 26
  Body mass measured in kilograms using a scale
Blood Pressure | Baseline, Week 12 and Week 26
  Systolic and Diastolic blood pressure
Triglyceride concentration | Baseline, Week 12 and Week 26
  From a blood sample
Low Density Lipids (LDL) concentration | Baseline, Week 12 and Week 26
  From a blood sample
Cholesterol concentration | Baseline, Week 12 and Week 26
  From a blood sample
Glucose concentration | Baseline, Week 12 and Week 26
  From a blood sample
HbA1c concentration | Baseline, Week 12 and Week 26
  From a blood sample
Patient Global Assessment of disease Impact | Baseline, week 8, week 12 and week 26
  Patient-reported degree of patient's perceived impact of their knee OA on their overall life will be obtained using a 100 mm analogue scale (VAS) with anchors: 0=" No impact" and 100 = "Worst imaginable impact".
Physical Functioning | Baseline, week 8, week 12 and week 26
  The Knee injury and Osteoarthritis Outcome Score (KOOS) function subscale (KOOS-function), a disease-specific patient-reported instrument designed to assess physical functioning in patients with knee osteoarthritis.
  The KOOS-function subscale is scored on a 0-100 scale with 100 indicating no functional impairments and 0 indicating extreme functional impairments.
Health related quality of Life and physical and mental well-being (Short Form 12 (SF-12)) | Baseline, week 8, week 12 and week 26
  The 12-item short form health questionnaire (SF-12) is a measure of physical and mental health.
  The physical health component is scored between 0-72. The mental health component is scored between 0-70. For both components 0 mean a worse outcome.

OTHER OUTCOMES:
Knee-related Quality of Life | Baseline, week 8, week 12 and week 26
  The Knee injury and Osteoarthritis Outcome Score (KOOS) quality of life subscale (KOOS-QoL), a disease-specific patient-reported instrument designed to assess knee-related quality of life in patients with knee osteoarthritis.
  The KOOS-QoL subscale is scored on a 0-100 scale with 100 indicating best possible knee-related quality of life and 0 indicating worst possible knee-related quality of life.
Knee Symptoms | Baseline, week 8, week 12 and week 26
  The Knee injury and Osteoarthritis Outcome Score (KOOS) symptoms subscale (KOOS-symptoms), a disease-specific patient-reported instrument designed to knee symptoms in patients with knee osteoarthritis.
  KOOS-symptom is scored on a 0-100 scale with indicating no symptoms and 0 indicating worst possible symptoms.
Knee Function in Sports and Recreational activities | Baseline, week 8, week 12 and week 26
  The Knee injury and Osteoarthritis Outcome Score (KOOS) Sports and Recreation subscale (KOOS-Sports/Recreation), a disease-specific patient-reported instrument designed to knee symptoms in patients with knee osteoarthritis.
  KOOS-Sports/Recreation is scored on a 0-100 scale with indicating no symptoms and 0 indicating worst possible symptoms.
The World Health Organisation - Five Well-Being Index (WHO-5) | Baseline, week 8, week 12 and week 26
  Patient reported mental well-being will be obtained with the The World Health Organisation 5-Well-Being Index consisting of five questions each scored on a 0 to 5 scale.
  Raw score: 0 represents worst possible well-being and 25 represents best possible well-being.
  Percentage score: 0 represents worst possible well-being and 100 represents best possible well-being.
OMERACT-OARSI treatment responder criteria | Baseline, week 8, week 12 and week 26
  A classification of patients as a positive responder based on the Outcome Measures in Rheumatology (OMERACT) and Osteoarthritis Research Society International (OARSI) (OMERACT-OARSI) responder criteria that classifies patients according to improvements in pain (co-primary outcome),function (secondary outcome) and patient global assessment (secondary outcome).
  Each participant is classified as either a "responder" or a "non-responder" at each of the post-baseline follow-ups.
Sleep quality using the global Single-item sleep quality scale (SQS) | Baseline, week 8, week 12 and week 26
  Sleep quality will be obtained with the global Single-item sleep quality scale (SQS). SQS is scored on 0-10 scale with 0 representing worst possible sleep quality and 10 representing best possible sleep quality.
Nightly pain | Baseline, week 8, week 12 and week 26
  Self-reported pain during the night is obtained on a 0-2 scale with 0=No nightly pain, 1=pain at movement or in certain positions, and 2=Pain even without movement.
Maximal aerobic capacity (VO2 peak) during a cardiopulmonary exercise test | Baseline, week 8, week 12 and week 26
  A cardiopulmonary exercise test will be used to assess maximal aerobic capacity (VO2peak) measured in ml/min/kg.
Maximum work during a cardiopulmonary exercise test | Baseline, week 8, week 12 and week 26
  The maximal work during the cardiopulmonary exercise test measured in Watts (W)
Respiratory exchange ratio (RER) during a cardiopulmonary exercise test | Baseline, week 8, week 12 and week 26
  The respiratory exchange ratio (RER) during the cardiopulmonary exercise test is calculated as the ratio of carbon-dioxide production (VCO2) and oxygen consumption (VO2)
Maximal hear rate during a cardiopulmonary exercise test | Baseline, week 8, week 12 and week 26
  The maximal heart rate during a cardiopulmonary exercise test is recorded as beats/min.
Lean body mass from a dual x-ray absorptiometry scan | Baseline, Week 12 and Week 26
  Dual x-ray absorptiometry (DXA) will be used to assess lean body mass
Total fat mass from a dual x-ray absorptiometry scan | Baseline, Week 12 and Week 26
  Dual x-ray absorptiometry (DXA) will be used to assess total fat mass.
Bone mineral density from a dual x-ray absorptiometry scan | Baseline, Week 12 and Week 26
  Dual x-ray absorptiometry (DXA) will be used to assess bone density.
Hip and waist circumstance | Baseline, Week 12 and Week 26
  The measurements are recorded in cm and measured during a clinical examination using a measurement tape and standardized procedures
Leg extensor power | Baseline, Week 12 and Week 26
  Muscle power (force × velocity) of the lower limb of the target knee will be assessed using the Nottingham power rig. In a seated position, the participants will be instructed to push with a single leg against a plate at maximal effort/force.
Analgesics usage | Baseline, Week 12 and Week 26
  The participants' use of over-the-counter paracetamol and ibuprofen will be recorded during an interview with an investigator.
Pressure pain sensitivity | Baseline, Week 12 and Week 26
  A hand-held pressure algometer will used to assess pressure pain thresholds (PPTs). Pressure will be applied at a rate of approximately 30 kilopascal per second (kPa/s), with a 1 cm2 probe. All participants are instructed to push a button when they feel that the pressure becomes just barely painful. PPTs from the medial tibiofemoral joint space on the target knee and the contralateral elbow will be assessed
C-reactive protein concentration | Baseline, Week 12 and Week 26
  From a blood sample
Interleukin 6 (IL6) concentration | Baseline, Week 12 and Week 26
  From a blood sample
Seismocardiography - estimate of maximal oxygen consumption (VO2max) during rest. | Baseline, Week 12 and Week 26
  Seismocardiography (SCG) is a technique for non-invasive evaluation of cardiac activity through the measurement of precordial vibrations using an accelerometer. SCG is performed by mounting a 3-axis accelerometer on the skin covering the sternum with double adhesive tape. The measurement is performed with the participant lying in the supine position after 5 minutes of rest. The 3-dimensional accelerations are recorded and used together with age, sex, body weight and height in an algorithm to estimate cardiorespiratory function (VO2max) at rest.
  NOTE: This outcome is added to the protocol after recruitment was started and will therefore only be measured on a subset of participants (participants enrolled after August 15, 2024).

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code